CLINICAL TRIAL: NCT04848363
Title: Analgesic Effect of Quadratus Lumborum Block in Laparoscopic Hemicolectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Evgenii Bespalov,MD, Doctor of the department of anesthesiology and resuscitation, Petrovsky National Research Centre of Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEK25011994
Record Dates: First submitted 2021-03-12; First posted 2021-04-19 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Distribution: randomized Intervention model: parallel distribution 2 groups
  * Control group: patients receiving general anesthesia with propofol, fentanyl and cisatracurium for induction and sevoflurane, fentanyl and cisatracurium for maintaining anesthesia. Patients receiving postoperative multimodal intravenous analgesia with paracetamol, ketoprofen, tramadol, and trimeperidine. Before surgery will be performde bilateral blockade of the QL muscle with normal saline.
  * Study group: patients receiving general anesthesia with propofol, fentanyl and cisatracurium for induction and sevoflurane, fentanyl and cisatracurium for maintaining anesthesia. Patients receiving postoperative multimodal intravenous analgesia with paracetamol, ketoprofen, tramadol, and trimeperidine. The QL blockade will be performed under ultrasound guidance using 20 ml of a solution of levobupivacaine 2.5 mg / ml.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blindness. The Principal Investigator performing the blockade knows the randomization group. The anesthesiologist, postoperative pain assessor, and study participant do not know the randomization group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): patients receiving general anesthesia with propofol, fentanyl and cisatracurium for induction and sevoflurane, fentanyl and cisatracurium for maintaining anesthesia. Patients receiving postoperative multimodal intravenous analgesia with paracetamol, ketoprofen, tramadol, and trimeperidine. In this group, after induction of anesthesia before the operation, bilateral blockade of the square dorsi muscle is performed under ultrasound guidance using 20 ml of a solution of levobupivacaine 2.5 mg / ml.
  Interventions: Procedure: Quadratus lumborum block
- Control group (Placebo Comparator): patients receiving general anesthesia with propofol, fentanyl and cisatracurium for induction and sevoflurane, fentanyl and cisatracurium for maintaining anesthesia. Patients receiving postoperative multimodal intravenous analgesia with paracetamol, ketoprofen, tramadol, and trimeperidine. In this group, after induction of anesthesia before surgery, bilateral blockade of the square dorsi muscle is performed under ultrasound guidance using 20 ml of saline.
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Quadratus lumborum block — QL block will be used for perioperative anesthesia. The blockade will be performed bilaterally by levobupivacaine (20ml) at concentration 0.25%.

SUMMARY:
Comparison of the effectiveness: Quadratus lumborum (QL) block by levobupivacaine with placebo.

DETAILED DESCRIPTION:
All patients will receive standard anaesthesia using fentanyl, protocol, cisatracurium and sevoflurane. Prevention of nausea and vomiting is performing using Apfel score.

All patients will receive post operative multimodal analgesia using paracetamol, ketoprofen, tramadol, and trimeperidine if numerical rating scale > 3 The study assumes use of QL block by levobupivacaine.in comparison with placebo in order to demonstrate the effectiveness of QL block during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone left-sided or right-sided laparoscopic hemicolectomy.
* Patient's willingness and ability to sign an informed consent document

Exclusion Criteria:

* Allergy to local anesthetics
* Chronic pain syndrome and associated opioid use.
* Coagulopathy
* Uncontrolled diabetes mellitus
* Physical Status Classification System scale above 3
* Diseases associated with the pathology of the hypothalamus
* Diseases associated with the pathology of the pituitary gland
* Diseases associated with the pathology of the adrenal glands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
NRS (Numeric rating scale) | two hours after surgery
  NRS scale 0-10, "no pain"; 10, "worst pain imaginable"

SECONDARY OUTCOMES:
The need for opioid analgesics during surgery | on operations
The need for opioid analgesics for postoperative pain relief | 72 hours after surgery
The need for antiemetic drugs to relieve postoperative nausea and vomiting | 12 hours after the surgery
Occurrence of prolonged post-operative ileus | first two weeks after surgery
Blood glucose level | after induction into anesthesia, immediately after the end of the surgery, 12 hours after the surgery
The level of blood lactate | after induction into anesthesia, immediately after the end of the surgery, 12 hours after the surgery
The level of cortisol in the blood | after induction into anesthesia and immediately after the end of the surgery
The level of prolactin in the blood | after induction into anesthesia and immediately after the end of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Petrovsky Research National Centre of Surgery ( Petrovsky NRCS), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
All patient data will be confidential